CLINICAL TRIAL: NCT01620437
Title: A Randomised, Double-blind, Single-centre, Two-Period Crossover Trial Testing the Bioequivalence of Two Formulations of NN-X14Mix50 in Healthy Japanese Subjects
Brief Title: Bioequivalence of Two Formulations of Biphasic Insulin Aspart 50 in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1581
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental)
  Interventions: Drug: biphasic insulin aspart 50
- Formulation B (Experimental)
  Interventions: Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — A single dose administrated subcutaneously (s.c., under the skin) on two separate dosing visits. A wash-out period of 6-21 days will take place between dosing visits

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the bioequivalence of two formulations of biphasic insulin aspart 50 (NN-X14Mix50) in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index) between 19-29 kg/m^2 (both inclusive)
* Fasting blood glucose between 3.8-6.0 mmol/L (both inclusive)
* Non-smokers

Exclusion Criteria:

* Subjects with a first-degree relative with diabetes mellitus
* Subjects smoke 5 cigarettes or more per day

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11-29 (Actual); Primary Completion 2003-12-30 (Actual); Study Completion 2003-12-30 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart curve in the interval from 0-16 hours
Cmax, maximum insulin aspart concentration

SECONDARY OUTCOMES:
tmax, time to maximum insulin aspart concentration
Area under the insulin aspart curve
Mean residence time (MRT)
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com